CLINICAL TRIAL: NCT01271127
Title: Screening for Coronary Artery Disease After Mediastinal Irradiation in Hodgkin Lymphoma Survivors
Brief Title: Screening for Coronary Artery Disease After Mediastinal Irradiation
Acronym: SCAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, L.A.Daniels, MD, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: NL31278.058.10
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Radiation Therapy; Coronary Artery Disease; Hodgkin Lymphoma
Keywords: radiation therapy; coronary artery disease; Hodgkin Lymphoma
MeSH Terms: conditions — Coronary Artery Disease; Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: CT coronary angiography — patient will undergo one CT coronary angiography

SUMMARY:
Survivors of Hodgkin Lymphoma (HL) are known to have an increased risk of developing late treatment sequelae such as cardiovascular events due to coronary artery disease. At present no active screening is performed in these patients since it is not known whether screening and subsequent treatment by means of revascularization is effective in reducing the risk of cardiovascular events in symptomatic individuals. In the trial the efficacy and therapeutic consequences of screening for coronary artery diasease by multi-slice CT (MSCT) among asymptomatic HL survivors will be evaluated.

DETAILED DESCRIPTION:
Objectives:

1. to determine whether MSCT as a screening method of HL survivors treated with mediastinal irradiation accurately identifies asymptomatic significant coronary artery disease.
2. to establish the prevelance of coronary abnormalities in HL survivors treated with mediastinal irradiation
3. to determine the frequency and type of intervention
4. to evaluate the acceptance of screening and asses quality of life among Hl survivors.

Study polulation:

50 long term survivors of HL, previously treatef with mediastinal irradiation without present evidence of cardiovascular disease

Intervention:

CT-coronary angiography and calcium score, to be performed as a screening method (to indicate further diagnostic treatent procedures)

ELIGIBILITY:
Inclusion Criteria:

* history of Hodgkin Lymphoma(all stages) with at least 10 disease free survival
* current age between 35-60
* mediastinal irradiation as part of HL treatment, radiotherapy data available
* written informed consent

Exclusion Criteria:

* current treatment for cardiovascualr disease, excelt hypertension hypercholesterolemia or cardiac murmurs
* known or sypmtomatic heart failure
* impaired kidney function (Cockcroft < 55 ml/min)
* known contrast allergy
* invasive angiography in past 2 years
* presence of life threatening disorder

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
accurately identifying asymptomatic coronary artery disease | one year
  to determine whether Ct coronary angiography as a screening method acuurately identifies asymptomatic coronary artery disease in a high risk poulation (HL survivors after mediastinal irradiation)

SECONDARY OUTCOMES:
prevalnce of cornary artery disease and frequency/type of subsequent intervention | one year
  to establish the prevelence of coronary abnormalities in HL survivors treated with mediastinal irradiation, and to determine the frequency and type of subsequent interventions

CONTACTS AND LOCATIONS:
Overall Officials: A.D.G. KRol, MD, PhD, Principal Investigator — Leiden University Medical Centre
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

REFERENCES:
- [Derived] Daniels LA, Krol SD, de Graaf MA, Scholte AJ, van 't Veer MB, Putter H, de Roos A, Schalij MJ, van de Poll-Franse LV, Creutzberg CL. Impact of cardiovascular counseling and screening in Hodgkin lymphoma survivors. Int J Radiat Oncol Biol Phys. 2014 Sep 1;90(1):164-71. doi: 10.1016/j.ijrobp.2014.05.038. PMID 25195991
- [Derived] Daniels LA, Krol AD, de Graaf MA, Scholte AJ, Van't Veer MB, Putter H, de Roos A, Schalij MJ, Creutzberg CL. Screening for coronary artery disease after mediastinal irradiation in Hodgkin lymphoma survivors: phase II study of indication and acceptancedagger. Ann Oncol. 2014 Jun;25(6):1198-203. doi: 10.1093/annonc/mdu130. Epub 2014 Mar 31. PMID 24692582